CLINICAL TRIAL: NCT01699451
Title: DNA, Blood and Skin Cell Repository for Research on ALS and Related Neurodegenerative Disorders at Mayo Clinic Florida
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bjorn E. Oskarsson, PI, Mayo Clinic
Other Study IDs: 12-004718
Record Dates: First submitted 2012-09-30; First posted 2012-10-03 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This study will establish a repository of stored DNA, RNA, monocyte, lymphocyte and skin fibroblast samples from people with ALS and ALS-FTD, subjects with a family history of ALS who do not have ALS or ALS-FTD, and subjects with no personal history of ALS or dementia, to support future translational and basic research studies on ALS and related neurodegenerative disorders.
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is intended to obtain clinical information and establish a repository of DNA, RNA, peripheral blood monocyte, lymphocyte and skin tissue samples from people with ALS and related neurodegenerative motor neuron diseases, people with a family history of these conditions, and healthy people with no family history of these disorders. The samples will be used in future research to learn about how these disorders affect people, what causes these conditions, and how the investigators can tell when someone has this kind of disease. Future research may also include the generation of stem cells from stored blood cell and skin cell samples. Participants will not be paid for taking part in this study.

ELIGIBILITY:
Inclusion Criteria:

* ALS Patient

  1. Clinical diagnosis of possible, laboratory-supported probable, probable or definite ALS according to modified EL Escorial criteria, suspected ALS according to original El Escorial criteria, or diagnosis of a neurodegenerative disorder with evidence of ALS plus extramotor features
  2. > or = 18 years of age and willing to provide consent, or assent, if unable to consent
* Subject with family history of ALS or other relevant neurodegenerative disease

  1. No personal history of ALS, ALS-FTD or other motor neuron disease
  2. Family history of ALS, ALS-FTD in a first, second or third degree blood relative
  3. > or = 18 years of age and willing to provide consent
* Control

  1. No personal or family history (first or second degree blood relative) of ALS, dementia, Parkinson disease or other relevant neurodegenerative disorder
  2. > or = 18 years of age and willing to provide consent

Exclusion Criteria:

* ALS Subject and subject with family history of ALS/ALS-FTD or other neurodegenerative motor neuron disorder but no personal history of such conditions

  1. History of medical disorder that leaves in question whether neurological signs and symptoms potentially related to a neurodegenerative disease may be contributed to by an acquired condition
  2. Limited mental capacity rendering the subject unable to comply with skin punch biopsy or standard phlebotomy procedures
  3. For collection of skin punch biopsy, an increased risk of bleeding complications or allergy to local anesthetic administered at the time of skin biopsy
* Healthy Control Subject

  1. Personal or family history of dementia or other neurodegenerative disease (Parkinson disease, Alzheimer disease, etc.)
  2. Limited mental capacity rendering the subject unable to provide written informed consent or comply with standard phlebotomy procedures
  3. For collection of skin punch biopsy, an increased risk of bleeding complications or allergy to local anesthetic administered at the time of skin biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be female or male, > or = 18 years of age. ALS and control subjects will meet eligibility criteria. Control subjects will be similar in age to ALS patients. No special classes of subjects are specifically sought or excluded from the protocol.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Repository sample collection | once

CONTACTS AND LOCATIONS:
Overall Officials: Bjorn Oskarsson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials